CLINICAL TRIAL: NCT06816472
Title: Evaluation of Leadership and Work Environment in the Process of Integrating Evidence-based Practices in Surgical Clinics: A Multicenter Study
Brief Title: Evidence-based Nursing Practice in Surgical Clinics
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: Evidence-based Practice
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Evidence Based Nursing; Leadership
Keywords: Evidence based nursing; Leadership; Woek environment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgical nurses: It will be carried out with nurses working in the surgical units of Aydın Adnan Menderes University Practice and Research Hospital, the City Hospital and Süleyman Demirel University Research and Practice Hospital in Isparta province and Burdur State Hospital in Burdur province (General Surgery, Urology, Orthopedics and Traumatology, ENT/Eye/Plastic and Reconstructive Surgery, Brain Surgery, Gynecology and Obstetrics, Pediatric Surgery and Day Surgery clinics, Surgical Intensive Care, General Intensive Care, Cardiovascular Intensive Care, Brain Surgery Intensive Care, Anesthesia Intensive Care, Emergency Service and Day Hospital, Operating Room Service).

SUMMARY:
It is aimed to examine the leadership status and work environments of nurses working in surgical units during the integration of evidence-based practices into the institution.

DETAILED DESCRIPTION:
The study will be conducted with 248 nurses working in surgical units of three centers in Aydın, Isparta and Burdur provinces. Before the data collection begins, nurses will be informed about the study. The study data will be collected by researchers through face-to-face interviews with nurses every weekday between 15:00-16:00, so that the daily operations of the nurses and the institution will not be affected. The purpose of the study will be explained to the nurses who will participate in the study and the nurses who volunteer to participate will be asked to fill out the form. The form will take approximately 15 minutes to fill out. The study will question the sociodemographic characteristics of the nurses, their leadership status in the process of integrating evidence-based practices into the clinic, and the work environment and influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Having worked in a surgical unit for at least six months

Exclusion Criteria:

* Not being a graduate of the nursing department

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It will be carried out in three centers in Aydın, Isparta and Burdur provinces with 248 nurses working in General Surgery, Urology, Orthopedics and Traumatology, ENT/Eye/Plastic and Reconstructive Surgery, Brain Surgery, Gynecology and Obstetrics, Pediatric Surgery and Day Surgery clinics, Surgical Intensive Care, General Intensive Care, Cardiovascular Intensive Care, Brain Surgery Intensive Care, Anesthesia Intensive Care, Emergency Service and Day Hospital, Operating Room Services.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Leadership in Evidence-Based Practice | Once between 01.10.2024 and 31.05.2025
  This is the first section of the scale and consists of 10 items. Scale items are scored using a 5-point Likert system ranging from 1 (strongly disagree) to 5 (strongly agree). A minimum of 10 and a maximum of 50 points are obtained from the scale. As the score obtained from the scale increases, it is interpreted that leadership in evidence-based practices increases.
Evidence-Based Practice Work Environment | Once between 01.10.2024 and 31.05.2025
  This is the second part of the scale and consists of 8 items. Scale items are scored using a 5-point Likert system ranging from 1 (strongly disagree) to 5 (strongly agree). A minimum of 8 and a maximum of 40 points are obtained from the scale. As the score obtained from the scale increases, it is interpreted that the working environment improves in evidence-based practices.

SECONDARY OUTCOMES:
Factors Affecting the Leadership and Work Environments of Surgical Nurses in the Process of Integration of Evidence-Based Practices into the Clinic | Once between 01.10.2024 and 31.05.2025
  The effects of nurses' sociodemographic characteristics on primary outcomes will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Arslan, PhD, Study Director — Director; Filiz Salman Saraç, PhD, Study Chair — Researcher; Hatice Ersoy, PhD, Study Chair — Researcher; Sultan Özkan, PhD, Study Chair — Researcher
Locations (1):
- Ezgi Arslan, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.